CLINICAL TRIAL: NCT03049774
Title: A Retrospective Study of the Recombinant Human Interleukin-11 (I) (Baijieyi) for Prevention and Treatment of Chemotherapy-induced Thrombocytopenia in Patients With Malignant Tumor
Brief Title: A Study of the Recombinant Human Interleukin-11 (I) (Baijieyi) for Prevention and Treatment of Chemotherapy-induced Thrombocytopenia in Patients With Malignant Tumor
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Angde Biotech Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: EY201608
Record Dates: First submitted 2017-01-23; First posted 2017-02-10 (Actual); Last update posted 2017-02-10 (Actual); Status verified 2016-08

CONDITIONS: Chemotherapy-induced Thrombocytopenia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this retrospective study is to review and describe the safety and the efficacy of recombinant human interleukin-11 (I) i (Baijieyi), using information already recorded in 20 medical records, The time periods include May 8th of 2008 to december 31st of 2016.

ELIGIBILITY:
Inclusion Criteria:

1. prescriptions explicitly given to the injection of Baijieyi;
2. confirmed by histopathological or cytological examination of malignant tumors and chemotherapy;
3. treatment: platelet count had reached below 75×10^9/L after the treatment of chemotherapy and before using Baijieyi; prevention: patients with chemotherapy at the beginning of the preventive administration of BaiJieyi, and chemotherapy is same with previous cycle;
4. male or female, aged 18-85 years;
5. The main research information required is complete.

Exclusion Criteria:

1. using other platelets of chemicals or biological products in the in the chemotherapy cycle used Baijieyi;
2. using drugs which can cause thrombocytopenia in the in the chemotherapy cycle used Baijieyi;
3. bone marrow dysfunction or bone marrow involvement;
4. There are other causes of thrombocytopenia, such as aplastic anemia, acute leukemia, radiation sickness, immune thrombocytopenic purpura, and hypersplenism, in the course of the use of Baijieyi.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 20 clinical centers: subjects.who have received one or more injections of Baijieyi for treatment or prevention of chemotherapy-induced thrombocytopenia
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2017-02-28 (Estimated); Primary Completion 2017-08 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Days that platelet count firstly rebound to 75×10^9/L, 100×10^9/L, respectively, from the first time below 75×10^9/L at the chemotherapy cycle and the last chemotherapy cycle | 56 days
  For prevention
Days that platelet count firstly rebound to 75×10^9/L, 100×10^9/L | 28 days after the administration of Baijieyi
  For treatment

SECONDARY OUTCOMES:
the maximum and minimum platelet count at the chemotherapy cycle and the last chemotherapy cycle | 56 days
  For prevention
the lasting days of platelet count below 50×10^9/L at the chemotherapy cycle and the last chemotherapy cycle | 56 days
  For prevention
The number of platelet transfusions at the chemotherapy cycle and the last chemotherapy cycle | 56 days
  For prevention
the percentage of patients whose platelet count firstly recovered above 75×10^9/L and 100×10^9/L | 28 days after the administration of Baijieyi
  For treatment
the maximum and minimum platelet count, the lasting days of platelet count below 50×10^9/L | 28 days after the administration of Baijieyi
  For treatment
The number of platelet transfusions | 28 days after the administration of Baijieyi
  For treatment

OTHER OUTCOMES:
adverse events, serious adverse events, laboratory tests, ECG | 28 days after the administration of Baijieyi

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China